CLINICAL TRIAL: NCT06774508
Title: The Feasibility of a High-intensity Functional Exercise Program with Simultaneous Cognitive Challenge to Improve Physical and Cognitive Function in Older People with Intermediate Risk for Falls: a Randomized Controlled Pilot Trial
Brief Title: Feasibility of High-intensity Functional Exercise with Simultaneous Cognitive Challenge for Older People with Falls Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Annika Toots, Associate professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr 2024-07683-01
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Accidental Falls; Postural Balance; Gait; Cognition
Keywords: Accidental falls; Postural balance; Gait; Cognition; Exercise therapy; Resistance training; Aged

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation. Participants will receive repeated instructions not to disclose their group allocation to the assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity functional exercise with cognitive challenge (HIFE+Cog) (Experimental): High intensity functional exercise (HIFE+Cog) program with simultaneous cognitive challenge, individually tailored and performed twice weekly for 12 weeks, in supervised groups.
  Interventions: Other: HIFE+cog
- High-intensity functional exercise (HIFE) (Active Comparator): High intensity functional exercise (HIFE) program, individually tailored and performed twice weekly for 12 weeks, in supervised groups.
  Interventions: Other: HIFE

INTERVENTIONS:
Other: HIFE+cog — Each session will consist of individually tailored exercises performed at weight- bearing positions and covering lower leg strengthening exercises, as well as static- and dynamic balance exercises. Simultaneous cognitive exercises are added to static and dynamic balance exercises. Relative exercise intensity is encouraged to be moderate to high, and progressively adjusted by for example altering load or difficulty of the exercise. Session duration is 1 hour, including warm-up.
  Arms: High-intensity functional exercise with cognitive challenge (HIFE+Cog)
Other: HIFE — Each session will consist of individually tailored exercises performed at weight- bearing positions and covering lower leg strengthening exercises, as well as static- and dynamic balance exercises. Relative exercises intensity is encouraged to be moderate to high, and progressively adjusted by for example altering load or difficulty of the exercise. Session duration is 1 hour, including warm-up.
  Arms: High-intensity functional exercise (HIFE)

SUMMARY:
This study aims to evaluate the feasibility of a high-intensity functional exercise program with simultaneous cognitive challenge (HIFE+cog) among older people at risk of falls. The evaluation design and intervention development will be assessed with the following specific aims:

1. To investigate the acceptability and safety of the HIFE+cog program in older people at risk of falls, and the methods used in the study by evaluating recruitment, compliance with the intervention, severity of adverse events reported, and participant experiences.
2. To measure key outcome variables, including completion rates, missing data, estimates, variances, and 95% confidence intervals for between-group differences.

The study is designed as a randomized controlled pilot trial. Eligible participants will be randomized to either the intervention group (HIFE+cog) or the active control group (HIFE) to partake in individually tailored exercise, supervised and progressed by a physiotherapist, two times per week for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* aged 75 years or older
* moderate risk of falling (feeling unsteady or afraid of falling, or having fallen in the past year, with a self-selected gait speed ≤0,8 m/s or TUG >15 s without walking aid)
* can walk independently indoors, without a walking aid
* can walk 500m independently outdoors, with or without a walking aid

Exclusion Criteria:

* a high fall risk (≥2 falls in the past year, serious injury e.g. hip fracture from a fall in the past year requiring medical care, or inability to get up from the floor after a fall)
* Mini-Mental State Examination (MMSE) score <24 or dementia diagnosis
* a medical condition that may affect participation in high-intensity gait, balance, and leg strength exercise, or other movement-related conditions affecting exercise or tests (e.g., pain, dizziness, visual or hearing impairment)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Before intervention start
  Rate of recruited participants, and sources for recruitment
Adherence | Through the 3-month intervention
  Number of exercise sessions attended
Exercise intervention content and delivery | Through the 3-month intervention
  Number of exercises, sets, repetitions, and intensity achieved measured using a standardized exercise diary completed by supervisors after each session
Retention | Through the 3-month intervention
  Number of participants that completed follow-ups
Safety | Through the 3-month intervention period
  Adverse events, including falls and discomfort reported during or between sessions by participants or supervisors, and measured using a standardized exercise diary completed by supervisors after each session
Balance and gait capacity | Baseline, 3 months
  The Timed up and go (TUG) test, with and without cognitive task
Balance and gait capacity | Baseline, 3 months
  The 4m forward gait speed test, with and without cognitive task
Balance and gait capacity | Baseline, 3 months
  The 4m backward gait speed test
Balance and gait capacity | Baseline, 3 months
  The Berg balance scale
Balance and gait capacity | Baseline, 3 months
  The 30-s Chair stand test
Cognitive function | Baseline, 3 months
  The Mindmore cognitive battery: Mental speed with The Symbol-Digit Processing test
Cognitive function | Baseline, 3 months
  The Mindmore cognitive battery: Mental speed with The Reaction test I and II
Cognitive function | Baseline, 3 months
  The Mindmore cognitive battery: Attention and executive function (shifting) with The Trail making test - Click (TMT-Click)
Cognitive function | Baseline, 3 months
  The Mindmore cognitive battery: Short term- and working memory with The Corsi Block test
Cognitive function | Baseline, 3 months
  The Mindmore cognitive battery: Executive function (inhibition) with The Stroop test
Cognitive function | Baseline, 3 months
  The Mindmore cognitive battery: Executive function (verbal fluency) with The FAS test
Occupational performance | Baseline, 3 months
  The Canadian Occupational Performance Measure (COPM)
Experiences of the intervention and effects | 3 months
  Individual interviews with participants in the intervention group

SECONDARY OUTCOMES:
Fear of falling | Baseline, 3 months
  The Falls Self-Efficacy Scale (FES-I)
Psychological wellbeing | Baseline, 3 months
  The Philadelphia Geriatric Center Morale Scale (PGCMS)
Physical activity | Baseline, 3 months
  The International Physical Activity Questionnaire-Elderly (IPAQ-E)
Depressive disorders | Baseline, 3 months
  The Geriatric Depression Scale (GDS-15)
Health related quality of life | Baseline, 3 months
  The EQ5D, Selected questions from The short form (36) Health survey
Activities of daily life (ADL) | Baseline, 3 months
  The Katz ADL Index
Descriptive information | Baseline
  Age, gender, education, living conditions, past and current medical conditions and medications from self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Annika Toots, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analysed during the study will not publicly available to protect the participants' confidentiality (in accordance with The General Data Protection Regulation, European Union Regulation) but are available from the principal investigator on reasonable request.